CLINICAL TRIAL: NCT06929871
Title: A Prospective Randomised Controlled Trial Comparing Cementless Mako Robotic-arm Assisted Total Knee Arthroplasty Versus Cemented Mako Robotic-arm Assisted Total Knee Arthroplasty.
Brief Title: Mako Cementless TKA vs Mako Cemented TKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151407
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Replacement; Total Knee Replacement Surgery; Total Knee Arthroplasty; Osteoarthritis (OA) of the Knee
Keywords: robotic surgery; cemented implants; uncemented implants; makoplasty; functional outcomes; clinical outcomes; radiological outcomes; inflammatory marker; radiostereometric analysis; RSA
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: prospective, randomised, single-site, single-blinded trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mako cementless TKA (Experimental): Mako robotic-arm assisted total knee arthroplasty using cementless implants
  Interventions: Device: Mako cementless TKA
- Mako cemented TKA (Active Comparator): Mako robotic-arm assisted total knee arthroplasty using cemented implants
  Interventions: Device: Mako cemented TKA

INTERVENTIONS:
Device: Mako cementless TKA — Mako robotic-arm assisted total knee arthroplasty using cementless implants
  Arms: Mako cementless TKA
Device: Mako cemented TKA — Mako robotic-arm assisted total knee arthroplasty using cemented implants
  Arms: Mako cemented TKA

SUMMARY:
The overall aims of this prospective, randomised, single-blinded controlled trial are to compare functional, radiological and clinical outcomes in Mako robotic-arm assisted cementless Total Knee Arthroplasty (TKA) versus Mako robotic-arm assisted cemented TKA.

DETAILED DESCRIPTION:
Osteoarthritis of the knee accounts approximately for 85% of the disease burden across the globe10. Almost one in six people is affected by knee arthritis and according to the latest National Joint Registry (NJR) report; over the last three years in England and Wales more than 100,000 patients underwent total knee replacement each year.

Registry-based studies have shown good clinical outcomes and survivorship following TKA, however despite these results aseptic loosening and lysis remain the leading indications for revision. Furthermore, there is a higher incidence of patient dissatisfaction compared to total hip arthroplasty, with up to 20% of patients reporting dissatisfaction in an otherwise uncomplicated TKA. There has been an exponential rise in the number of TKAs performed in the UK and around the world, with a sharp increase in the percentage of younger patients undergoing TKA11. Notwithstanding, younger patients have consistently shown poorer outcomes following TKAs and younger age has been recognised as a risk factor of aseptic loosening; thus raising a concern given the demographic trend of younger patients seeking TKA.

The optimal component fixation mode has been contentious, and it is yet to be established whether one is superior to the other. Early reports of cementless TKAs had risen concerns in relation to suboptimal fixation and early failure. However, since then, there has been a dramatic improvement in the design and technique of cementless TKA, reflected on several studies reporting promising and favourable outcomes with cementless fixation; a recent systematic review and meta-analysis has shown a 96% - 100% survival at ten- to 15-years. Proponents of the technique highlight the potential of biologic fixation and better osseointegration, given highly porous surfaces on TKA designs prevent a mismatch in stiffness and approximate the pore size and elasticity of trabecular bone. Moreover, cementless implants do not produce cement debris, averting the risk of cement degradation leading to prosthesis loosening. Commonly, cementless prostheses are more expensive than cemented, however a recent study reported a lower overall cost associated with cementless TKA; showing that the additional cost could be offset when additional variables are taken into account such as operating time, implant, cement and cementing accessories.

The evolution of surgical technology has led to the development of robotic-arm assisted TKA, which uses three dimensional images of each patient's unique anatomy to guide bone resection, implant positioning, and optimise limb alignment. The robotic arm interactive orthopaedic (RIO) system (Mako surgical) uses preoperative computerised tomography scans to build a computer-aided design (CAD) model of the patient's knee joint. The Mako robotic software processes this information to calculate the volume of bone requiring resection and creates a three-dimensional haptic window for the robotic arm to resect. The robotic arm has tactile and audio feedback to resect bone to a high degree of accuracy and preserve as much bone stock as possible. The surgeon can then plan and execute optimal sizing and positioning of the prosthesis to achieve the required bone coverage, minimise bone resection, and obtain the desired limb alignment. The Mako software also creates a patient-specific computer aided design model using the preoperative CT scan, which means that only bone anatomy is segmented. The surgeon is able to compensate for wear when creating the surgical alignment plan and uses intraoperative bone registration to map the patient's anatomy.

There are very few randomised prospective studies exploring clinical and radiological outcomes in cemented versus uncemented TKA. Prospective studies comparing functional outcomes between the treatment groups have been performed but the main limitation of these studies has been the inability to achieve the implant position to a high degree of accuracy. Furthermore, there is a paucity of long-term studies and limited data correlating radiological outcomes to clinical findings.

Since its introduction in 1974, radiostereometric analysis (RSA) has been widely used in the assessment of implant stability and survivorship in joint arthroplasty. The model-based RSA technique involves the insertion of inert tantalum beads into the bone around the prosthesis. These bone markers act as fixed reference points from which the spatial resolution and rotation of the implants are calculated. Early implant migration as assessed by RSA has been shown to accurately reflect the risk of loosening.

The most recent data comes from Hasan et al that conducted a RCT comparing the cementless Tritanium 3D-printed Tritanium TKA with its cemented counterpart using RSA and clinical outcomes. Authors reported a larger migration of the cementless TKA in the first three months, after which stabilisation was noted in in all cases with the exception of one malaligned TKA that was revised early. No intraoperative navigation or robotic systems were used, therefore weakening reproducibility of implant positioning.

While there have been RCTs comparing cemented to cementless TKA, there is no published study comparing these two groups utilising robotic-arm assistance, which is one of the fastest growing procedures in TKA. Cementless TKA is growing exponentially along with robotic TKA and it would be valuable to ascertain whether there is an advantage of cementless vs cemented TKA.

With the altering demographics of TKA, it is projected that by 2030, 55% of the patients pursuing TKA will be younger than 65 years old. There is a need for high quality evidence on the radiological and clinical benefits of cementless TKA compared to cemented TKA. It is possible to improve on previous studies by incorporating RSA, assessing implant migration and calculating the risk of early implant failure. Our study will also be characterised by high validity; recording a more comprehensive range of clinical and functional outcome measures, blinding patients and using long follow-up times. Furthermore, Mako robotic-arm assistance will be used to improve accuracy of bone resection, guide implant positioning, reduce soft tissue injury, and provide intraoperative assessment of limb alignment; therefore, minimising bias related to surgical variability and inconsistent implant positioning. Findings of this study will enable an improved understanding of the radiological, clinical and functional benefits of cementless fixation compared to cemented fixation in TKA. Findings of the trial could also be used to improve outcomes in total knee arthroplasty; better patient functional outcomes and satisfaction; improved cost-effectiveness by reducing operating time and cement cost; improved long-term implant survival; better outcomes for the exponentially growing number of younger patients pursuing TKA.

The overall aims of this prospective, randomised single-blinded controlled trial are to compare functional, radiological and clinical outcomes in Mako robotic-arm assisted cementless TKA (cementless TKA) versus Mako robotic-arm assisted cemented TKA (cemented TKA). Patients undergoing cemented TKA will form the control group and those undergoing cementless TKA will form the investigation group. A superiority trial design will be used to evaluate whether cementless TKA provides superior outcomes compared to cemented TKA. Radiostereometric analysis (RSA) will be used to assess differences in early and late implant migration between cementless TKA and cemented TKA.

The primary objective of this study is to compare Forgotten Joint score (FJS) at one year following surgery.

This study is a prospective, single-centre, randomised, single-blinded, controlled study. Patients undergoing cemented functionally aligned TKA will form the control group and those undergoing the cementless functionally aligned TKA will form the investigation group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has symptomatic knee osteoarthritis requiring primary TKA
2. Patient and surgeon are in agreement that TKA is the most appropriate treatment
3. Patient is fit for surgical intervention following review by surgeon and anaesthetist
4. Patient is over 18 years old at time of surgery
5. Gender: male and female
6. Patient must be capable of giving informed consent and agree to comply with the postoperative review program
7. Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

1. Patient is not suitable for routine primary TKA e.g. patient has ligament deficiency that requires a constrained prosthesis
2. Patient has bone loss that requires augmentation
3. Patient is not medically fit for surgical intervention
4. Patient requires revision surgery following previously failed correctional osteotomy or ipsilateral TKA
5. Patient has a DEXA scan with T-score < -2.5 at any point
6. Patient is immobile or has another neurological condition affecting musculoskeletal function
7. Patient is less than 18 years at time of surgery
8. Patient is unable or unwilling to sign the informed consent form specific to this study
9. Patient is unable to attend the follow-up programme
10. Previous pathological fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
The Forgotten Joint Score [FJS] | At one year post-op
  The Forgotten Joint Score (FJS) is a patient-reported outcome measure (PROM) used to assess the degree to which patients have "forgotten" their artificial joint, particularly after joint replacement surgery, like knee replacements.
  The score [100 is best] was developed to measure the success of a joint replacement by evaluating how well a patient has adjusted to the implanted joint in their daily life. It aims to show whether the patient feels like the artificial joint is part of their body and doesn't think about it in normal activities.
  The FJS has a series of questions about:
  * Pain or discomfort in the joint
  * Function and mobility
  * The awareness of the joint during daily activities (e.g., walking, climbing stairs, or sitting)
  * The patient's satisfaction with the joint. A high score means the patient feels that the joint replacement is functioning well and does not interfere with their quality of life, while a lower score may indicate that the patient is not fully satisfied.

SECONDARY OUTCOMES:
Assessement of tibial implant migration by maximum total point motion [MTPM] in millimetres using Radiostereometric analysis (RSA) | 1, 2 and 5-years post-op
  Radiostereometric analysis (RSA) is a highly precise imaging technique used in orthopedic research and clinical practice to track the movement of bones and implants within the body. It uses X-ray images taken from two different angles to create a 3D model of the bones or implants, which allows for highly accurate measurements of their position and motion over time. RSA is particularly useful for evaluating implant movement. It assesses the stability of orthopedic implants - for this outcome the tibial component of the knee prosthesis - to determine if it is moving, which could lead to failure. This study will assess continuous migration between the first and second year post-op, and second and fifth year post-op, measured by maximum total point motion [MTPM]: the maximum displacement observed between two objects (like a bone and an implant, or between two parts of an implant). Measurements are in millimetres [mm]; lower mm is better than higher mm, which could indicate loosening
Assess risk of loosening of the knee prosthesis by maximum total point motion [MTPM] in millimetres using Radiostereometric analysis [RSA] | 1, 2 and 5-years post-op
  Radiostereometric analysis [RSA] is a highly precise and advanced imaging technique used in orthopedic research and clinical practice to track the movement of bones and implants within the body. It uses X-ray images taken from two different angles to create a 3D model of the bones or implants, which allows for highly accurate measurements of their position and motion over time.
  RSA is particularly useful for evaluating implant movement. It assesses the stability of orthopedic implants - for this study the knee prosthesis - to determine if it is moving or loosening, which could lead to failure.
  This study will assess continuous migration between the first and second year pos-op, and second and fifth year post-op, measured by maximum total point motion [MTPM]: the maximum displacement observed between two objects (like a bone and an implant, or between two parts of an implant). Measurements are in millimetres [mm]; lower mm is better than higher mm, which could indicate loosening
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Preoperatively and postoperatively at 1 year, 2 years and 5 years
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used set of questionnaires designed to assess the severity of symptoms in patients, particularly in the knee and hip joints. For this study it is the knee joint It evaluates three main areas:
  Pain: How much pain the person experiences in their joints. Stiffness: How stiff the person feels in their joints. Physical Function: The difficulty the person has with everyday movements and activities.
  The WOMAC score is typically measured using a series of questions related to each of these areas, with responses indicating the level of severity. Each section is scored on a scale, and the total score is used to assess the degree of impact of their affect joint in their everyday life.
  The higher score the worse, the lower score the better outcome: 0 is the best score indicating no problems with pain, stiffness or physical function
The Oxford Knee Score (OKS) | Preoperatively and postoperatively at 1 year, 2 years and 5 years
  The Oxford Knee Score (OKS) is a patient completed questionnaire and assesses apatient's knee function and the severity of symptoms related to knee problems, particularly after knee surgery, such as knee replacement.
  The OKS consists of 12 questions related to symptoms, pain, and functional limitations. The questions focus on pain intensity, stiffness, and the ability to perform activities like walking, climbing stairs, and getting in and out of a car. Patients respond to each question on a 5-point scale, where higher scores generally indicate better knee function and less discomfort.
  The total score ranges from 0 to 48, with lower scores indicating more severe knee problems and higher scores indicating less pain and better function.
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | 1, 2 and 5-years post-op
  European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) is a tool used to measure a person's health-related quality of life. It assesses the impact of health conditions and treatments on a person's well-being.
  There are 2 parts:
  First part includes five dimensions:
  * Mobility
  * Self-care
  * Usual activities
  * Pain/discomfort
  * Anxiety/depression
  For each of these dimensions, the person selects one of three levels:
  * No problems
  * Some problems
  * Severe problems Second part: EQ-5D Visual Analog Scale (VAS): This is a self-rated scale where the person rates their overall health from 0 (worst imaginable health) to 100 (best imaginable health).
  The responses from the descriptive system can also be used to calculate a utility score. '1' is a perfect score, with anything from 0.99 and below a lesser score.
Analgesia requirements | Up to 90 days; also 1 year and 2 years
  Analgesic medication use: the type and frequency of use of analgesia
Mobility of knee joint | Up to 90 days; also 1 year and 2 years
  Range of movement (degrees) of knee joint measured with a goniometer of patient's full knee extension to full knee flexion. Knee extension of >10 degrees and knee flexion of <90 degrees would be a worse outcome; knee extension <10 degrees and knee flexion >90 degrees would be a better outcome
Length of operation | During operation/surgery
  Operating time (minutes)
Length of stay | Up to 90 days
  Time to discharge [minutes]; fewer minutes indicate better outcome
Preservation of posterior offset by measurement in millimetres of thickness of posterior condyle of the femur | Pre-operative and day 1 postoperative
  Measurement of maximum thickness of the posterior condyle projected posteriorly to the tangent of the posterior cortex of the femoral shaft on true lateral radiographs of the knee
Preservation of anterior offset by measurement in millimetres of anterior condyle height and the anterior offset index of the femur | Pre-operative and day 1 post-operative
  Measurement in millimetres of the anterior condylar height and the anterior offset index to assess the anterior projection of the femoral condyles.
Complications | Through study completion over 5 years
  Record any complication as well as need for further surgery. Fewer complications indicate better outcome
Assess systemic inflammatory reaction incited by cemented or cementless fixation | 1 week postoperatively
  Level of serum inflammatory cytokine in picograms per mililitre [pg/ml]: Interleukin-6 [IL-6]
Assess systemic inflammatory reaction incited by cemented or cementless fixation | 1 week postoperatively
  Level of serum inflammatory cytokine in picograms per mililitre [pg/ml]: Tumour necrosis factor-alpha [TNFa]
Assess systemic inflammatory reaction incited by cemented or cementless fixation | 1 week postoperatively
  Level of serum inflammatory cytokine in picograms per mililitre [pg/ml]: Erythrocyte Sedimentation Rate [ESR]
Assess systemic inflammatory reaction incited by cemented or cementless fixation | 1 week postoperatively
  Level of serum inflammatory cytokine in picograms per mililitre [pg/ml]: C-reactive protein [CRP]
Assess systemic inflammatory reaction incited by cemented or cementless fixation | 1 week postoperatively
  Level of serum inflammatory cytokine in picograms per mililitre [pg/ml]: Creatinine Kinase [CK]
Operating time costs in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Operating time and the cost in pounds sterling. Fewer pounds sterling indicates better outcome
Inpatient rehabilitation costs in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Inpatient rehabilitation and the costs in pounds sterling. Fewer pounds sterling indicates better outcome
Equipment and sterilisation costs in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Equipment and sterilisation and the costs in pounds sterling. Fewer pounds sterling indicates better outcome
Outpatient rehabilitation costs in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Outpatient rehabilitation and the costs in pounds sterling. Fewer pounds sterling indicates better outcome
Additional imaging costs - plain x-ray - in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Additional imaging costs of plain x-ray in pounds sterling. Fewer pounds sterling indicates better outcome
Additional imaging costs - CT scan - in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Additional imaging costs of CT scan in pounds sterling. Fewer pounds sterling indicates better outcome
Additional imaging costs - ultrasound scan - in pounds sterling | Through study completion over 5 years
  Comparisons between the two treatment groups relating to: Additional imaging costs of ultrasound scan in pounds sterling. Fewer pounds sterling indicates better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Fares S Haddad, MBBS MD (Res) MCh (Orth) FRCS, Study Chair — UCL Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No